CLINICAL TRIAL: NCT05011474
Title: Safety and Efficacy Study of Matrilin-3 Pretreated Autologous Adipose Derived Mesenchymal Stem Cells Implantation in Chronic Low Back Pain Patients With Lumbar Intervertebral Disc Degeneration
Acronym: MANT3_ASC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inbo Han (Other)
Responsible Party: Sponsor-Investigator, Inbo Han, Professor, Spine Neurosurgeon, Bundang CHA Hospital, CHA University
Organization: CHA University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10-013
Record Dates: First submitted 2021-08-17; First posted 2021-08-18 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Patients With Chronic Low Back Pain Due to Degenerative Lumbar Disc

STUDY DESIGN:
Intervention Model Description: This clinical trial is a Phase 1/2a, open and researcher-led clinical trial. Subjects will be enrolled in succession, signed informed consent, and administered an autologous adipose-derived mesenchymal stem cell spheroid pretreated with matrillin 3 to each eligible subject meeting all selection criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: administered an autologous adipose-derived mesenchymal stem cell spheroid pretreated with matrillin 3 — Adipose-derived mesenchymal stem cells isolated from subject's adipose tissue are pretreated with matrillin 3 and produced in spheroid form.

SUMMARY:
To investigate the safety and efficacy of autologous adipose-derived mesenchymal stem cell spheroids pretreated with matrillin-3 in chronic low back pain patients with lumbar intervertebral disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 19-70 years
* Among the subjects with low back pain, conventional conservative treatment is performed, but the back pain or hip pain persists for more than 3 months, and it is determined that the cause of the back pain is a degenerative disc (MRI checks for a degenerative disc)
* Has Oswestry Disability score(ODI) ≥ 30%
* Has Visual Analogue Scale(VAS) ≥ 4
* Between lumbar 1-sacral 1, Magnetic Resonance Imaging (MRI) grade according to the Pfirrmann classification is 3~4.
* Has one or two degenerative lumbar discs identified by MRI (Confirmation of low back pain due to disc through various nerve block procedures.)
* Consent was prepared for stem cell administration

Exclusion Criteria:

* Patient requiring surgery due to severe pain in lower extremities due to severe nerve compression due to severe lumbar stenosis or prolapse of lumbar nucleus.
* patient with spinal instability, spondylitis, or vertebral fracture
* type 3 Modic change is in an endplate
* Patient whose disc height has decreased by more than 1/2 due to severe disc degenerative change
* Patient with severe osteoporosis (The average value of the T score in the lumbar spine bone density test is -2.5 or less)
* has undergone surgery, such as disc resection, on the disc to which the cells will be administered
* Patient who received lumbar epidural steroid injection 3 weeks before cell administration
* Pregnant or lactating women
* Among female patients who are likely to become pregnant during the clinical trial, who do not use medically acceptable methods of contraception

  * medically acceptable methods of contraception: condom, Oral contraception lasting for at least 3 months, Has received an infusion pill before 3 months, using an injectable or implantable contraceptive, or installed an intrauterine contraceptive device
* has a history of psychiatry or who are currently undergoing treatment, who judged that it is difficult to proceed with the clinical trial under the judgment of the researcher
* Patient with drug or alcohol addiction who cannot understand the purpose and method of this clinical trial
* Patient who participated in other clinical trials within 3 months prior to participation in the trial
* Patient who may affect this clinical trial due to serious medical conditions (hypertension not controlled by drugs, diabetes not controlled by drugs, cirrhosis, kidney failure, tumors)
* Patient with a history of malignant tumors within the last 5 years
* has a history of administration of cell therapy products
* Other persons who have clinically significant findings deemed inappropriate for this clinical trial due to medical judgment by the person in charge of the clinical trial

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1) Adverse reaction and serious adverse reaction evaluation 2) laboratory inspection 3) Vital signs 4) Biochemical examination 5) Lumbar MRI 6) Monitoring systemic infection | During Clinical Trial Period
  It will be considered safe and tolerated in the absence of the following:
  * Grade 3 (NCI grading system) or higher adverse reactions related to cell products
  * Any evidence that the cells are contaminated with infectious substances
  * Any evidence that cells show tumorigenic potential

SECONDARY OUTCOMES:
Confirmation of the degree of pain improvement in VAS | before and at 1 week, 1, 3, 6 months after stem cell injection
  on a scale of 0 to 10, with 0 meaning no pain and 10 meaning the worst pain you can imagine
Confirmation of the degree of improvement in disability (ODI) | before stem cell injection and at 1 week, 1, 3, and 6 months after injection
  on a scale of 0 to 3, with 0 meaning no disability and 10 meaning severe disability
Confirmation of increase in water content in the nucleus using MRI | before stem cell injection and at 1 and 6 month after injection

CONTACTS AND LOCATIONS:
Locations (1):
- CHA University, CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://sites.google.com/view/inbolab/home